CLINICAL TRIAL: NCT05302414
Title: The Learning Outcome of Resuscitation Teamwork Training on Developing Teamwork Performance in Postgraduate Year Doctors and Nurses - Comparison of Board Game-based Learning, Simulation-based Learning and Lecture-based Learning.
Brief Title: The Learning Outcome of Resuscitation Teamwork Training in Postgraduate Year Doctors and Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N202201126
Record Dates: First submitted 2022-03-09; First posted 2022-03-31 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2022-08

CONDITIONS: Patient Care Team
Keywords: Teamwork; Resuscitation; Team training
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: three arms
Who Masked: Outcomes Assessor
Masking Description: two assessors using video to evaluate outcomes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Board game-based learning (experience group-I) (Experimental): The team of PGY doctors and nurses receive training in resuscitation teamwork skills through a board game-based teaching approach.
  Interventions: Behavioral: Board game-based learning
- Simulation-based learning (experience group-II) (Experimental): The team of PGY doctors and nurses receive training in resuscitation teamwork skills through a simulation-based teaching approach.
  Interventions: Behavioral: Simulation-based learning
- Lecture-based learning (control group) (Other): The team of PGY doctors and nurses receive training in resuscitation teamwork skills through an interactive lecture-based learning approach.
  Interventions: Behavioral: Lecture-based learning

INTERVENTIONS:
Behavioral: Board game-based learning — The team of PGY doctors and nurses received 3 hours training intervention in resuscitation teamwork skills through a board game-based teaching approach.
  Other Names: experience group-I
  Arms: Board game-based learning (experience group-I)
Behavioral: Simulation-based learning — The team of PGY doctors and nurses received 3 hours training intervention in resuscitation teamwork skills through a simulation-based teaching approach.
  Other Names: experience group-II
  Arms: Simulation-based learning (experience group-II)
Behavioral: Lecture-based learning — The team of PGY doctors and nurses received 3 hours training intervention in resuscitation teamwork skills through an interactive lecture-based approach.
  Other Names: control group
  Arms: Lecture-based learning (control group)

SUMMARY:
It is challenging for healthcare team to manage emergency patient effectively. Most of these critical patients have medical conditions and need complex medical managements. Research findings have shown that poor healthcare teamwork would result in poor communication, missing information, and insufficient situation monitoring and thus compromise patient safety. Simulation has been proved as an effective method to develop teamwork competency. However, comparing to traditional training model, simulation requires more resources such as funding, spaces, time, administration staffs, schedule, facilitators, and equipment. It would not be easy to delivery in various professional departments. Game-based learning was a known effective and learner-centered learning model which required less resources. Researchers have shown that game-based learning has higher acceptance for the learners and can improve learners' knowledge, attitude, motivation, and performance. Therefore, the aim of this study was to explore the learning effectiveness of resuscitation teamwork training of board game-based learning, simulation-based learning and lecture-based learning in PGY doctors and nurses.

DETAILED DESCRIPTION:
This will be a prospective, longitudinal, and randomized controlled trial design. A total number of 180 PGY doctors and nurses will be enrolled from a teaching hospital in northern Taipei City. They will be randomized into board game-based learning group, simulation-based learning group, and lecture-based learning group. Three groups will receive "Emergency Medical Response Teamwork" training and all of these contents were developed according to America Heart Association Guidelines for Cardiopulmonary Resuscitation and ECC and TeamSTEPPS curriculum from Agency for Healthcare Research and Quality. We will collect the professional demography, the professional medical knowledge for medical management, the concept of knowledge for teamwork, team performance, team attitude, medical management, course survey, and cognitive load scales. We will compare the learning effectiveness between three groups in pretest, posttest, and three-months follow up. Statistical methods used included descriptive and inferential statistics, χ2 chi-square tests, Kruskal-Wallis H test, Friedman test, Wilcoxon test, generalized estimating equations, and text mining.

ELIGIBILITY:
Inclusion Criteria:

1. Postgraduate Year doctors who is 20 years old and work in primary care.
2. Postgraduate Year nurses who is 20 years old and work in primary care

Exclusion Criteria:

1. Participant do not work in primary care provide.
2. Healthcare provider do not delivery in relative adult care department, such as pediatric department, obstetrics department, and psychiatry department so on.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-08-07 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Chieh Wu, Study Chair — Taipei Medical University Hospital
Locations (1):
- Jen-Chieh Wu, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboalshamat K, Khayat A, Halwani R, Bitan A, Alansari R. The effects of gamification on antimicrobial resistance knowledge and its relationship to dentistry in Saudi Arabia: a randomized controlled trial. BMC Public Health. 2020 May 13;20(1):680. doi: 10.1186/s12889-020-08806-2. PMID 32404076
- [Background] Al-Ghareeb AZ, Cooper SJ. Barriers and enablers to the use of high-fidelity patient simulation manikins in nurse education: an integrative review. Nurse Educ Today. 2016 Jan;36:281-6. doi: 10.1016/j.nedt.2015.08.005. Epub 2015 Aug 19. PMID 26323885
- [Background] Buijs-Spanjers KR, Harmsen A, Hegge HH, Spook JE, de Rooij SE, Jaarsma DADC. The influence of a serious game's narrative on students' attitudes and learning experiences regarding delirium: an interview study. BMC Med Educ. 2020 Sep 1;20(1):289. doi: 10.1186/s12909-020-02210-5. PMID 32873285
- [Background] Capella J, Smith S, Philp A, Putnam T, Gilbert C, Fry W, Harvey E, Wright A, Henderson K, Baker D, Ranson S, Remine S. Teamwork training improves the clinical care of trauma patients. J Surg Educ. 2010 Nov-Dec;67(6):439-43. doi: 10.1016/j.jsurg.2010.06.006. Epub 2010 Nov 5. PMID 21156305
- [Background] Fernandez R, Kozlowski SW, Shapiro MJ, Salas E. Toward a definition of teamwork in emergency medicine. Acad Emerg Med. 2008 Nov;15(11):1104-12. doi: 10.1111/j.1553-2712.2008.00250.x. Epub 2008 Oct 1. PMID 18828831
- [Background] Eddy K, Jordan Z, Stephenson M. Health professionals' experience of teamwork education in acute hospital settings: a systematic review of qualitative literature. JBI Database System Rev Implement Rep. 2016 Apr;14(4):96-137. doi: 10.11124/JBISRIR-2016-1843. PMID 27532314
- [Background] Cutumisu M, Patel SD, Brown MRG, Fray C, von Hauff P, Jeffery T, Schmolzer GM. RETAIN: A Board Game That Improves Neonatal Resuscitation Knowledge Retention. Front Pediatr. 2019 Jan 31;7:13. doi: 10.3389/fped.2019.00013. eCollection 2019. PMID 30766862
- [Background] Malmstrom B, Nohlert E, Ewald U, Widarsson M. Simulation-based team training improved the self-assessed ability of physicians, nurses and midwives to perform neonatal resuscitation. Acta Paediatr. 2017 Aug;106(8):1273-1279. doi: 10.1111/apa.13861. Epub 2017 May 3. PMID 28370414
- [Background] McEwan D, Ruissen GR, Eys MA, Zumbo BD, Beauchamp MR. The Effectiveness of Teamwork Training on Teamwork Behaviors and Team Performance: A Systematic Review and Meta-Analysis of Controlled Interventions. PLoS One. 2017 Jan 13;12(1):e0169604. doi: 10.1371/journal.pone.0169604. eCollection 2017. PMID 28085922
- [Background] Finer NN, Rich W. Neonatal resuscitation: toward improved performance. Resuscitation. 2002 Apr;53(1):47-51. doi: 10.1016/s0300-9572(01)00494-4. PMID 11947979
- [Background] Monsieurs KG, Nolan JP, Bossaert LL, Greif R, Maconochie IK, Nikolaou NI, Perkins GD, Soar J, Truhlar A, Wyllie J, Zideman DA; ERC Guidelines 2015 Writing Group. European Resuscitation Council Guidelines for Resuscitation 2015: Section 1. Executive summary. Resuscitation. 2015 Oct;95:1-80. doi: 10.1016/j.resuscitation.2015.07.038. Epub 2015 Oct 15. No abstract available. PMID 26477410
- [Background] Rosqvist E, Lauritsalo S, Paloneva J. Short 2-H in Situ Trauma Team Simulation Training Effectively Improves Non-Technical Skills of Hospital Trauma Teams. Scand J Surg. 2019 Jun;108(2):117-123. doi: 10.1177/1457496918789006. Epub 2018 Jul 20. PMID 30027817
- [Background] Sawyer T, Laubach VA, Hudak J, Yamamura K, Pocrnich A. Improvements in teamwork during neonatal resuscitation after interprofessional TeamSTEPPS training. Neonatal Netw. 2013 Jan-Feb;32(1):26-33. doi: 10.1891/0730-0832.32.1.26. PMID 23318204
- [Background] Truta TS, Boeriu CM, Copotoiu SM, Petrisor M, Turucz E, Vatau D, Lazarovici M. Improving nontechnical skills of an interprofessional emergency medical team through a one day crisis resource management training. Medicine (Baltimore). 2018 Aug;97(32):e11828. doi: 10.1097/MD.0000000000011828. PMID 30095658

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The total number of participants was 124, with 28 did not complete the pretest, resulting in 96 people completed pretest, intervention and posttest. Subsequently, 48 participants did not complete three-months follow up test , the total number of participants who completed the whole course reduced to 48.
Groups:
- Board Game-based Learning: The team of PGY doctors and nurses received training in resuscitation teamwork skills through a board game-based teaching approach.
- Simulation-based Learning: The team of PGY doctors and nurses received training in resuscitation teamwork skills through a simulation-based teaching approach.
- Lecture-based Learning: The team of PGY doctors and nurses received training in resuscitation teamwork skills through an interactive lecture-based learning approach.
Period: Pretest to Posttest
Arm/Group | Board Game-based Learning | Simulation-based Learning | Lecture-based Learning
Started | 44 | 40 | 40
Completed | 32 | 32 | 32
Not Completed | 12 | 8 | 8
Not completed — Lost to Follow-up | 12 | 8 | 8
Period: Posttest to Three Months Follow-up
Arm/Group | Board Game-based Learning | Simulation-based Learning | Lecture-based Learning
Started | 32 | 32 | 32
Completed | 16 | 16 | 16
Not Completed | 16 | 16 | 16
Not completed — Lost to Follow-up | 16 | 16 | 16

BASELINE CHARACTERISTICS:
Groups:
- Board-game Based Learning: The team of PGY doctors and nurses received training in resuscitation teamwork skills through a board game-based teaching approach.
- Total: Total of all reporting groups
Arm/Group | Board-game Based Learning | Simulation-based Learning | Lecture-based Learning | Total
Number analyzed (Participants) | 32 | 32 | 32 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.63 (4.16) | 24.31 (2.49) | 24.97 (3.04) | 24.97 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 24 | 77
  Male | 6 | 5 | 8 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 32 | 32 | 32 | 96
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Working experience (months) [Count of Participants; unit: Participants]
  0-6 months | 6 | 15 | 13 | 34
  7-12 months | 11 | 13 | 11 | 35
  13-18 months | 7 | 2 | 4 | 13
  19-24 months | 8 | 2 | 4 | 14
Education [Count of Participants; unit: Participants]
  Associate or below | 2 | 1 | 1 | 4
  Bachelor or above | 30 | 31 | 31 | 92
Units [Count of Participants; unit: Participants]
  Medical Ward | 4 | 8 | 6 | 18
  Surgical Ward | 9 | 2 | 7 | 18
  Special Unit | 8 | 8 | 2 | 18
  Operating Room | 3 | 9 | 10 | 22
  Others | 8 | 5 | 7 | 20
Resuscitation experience (times after work) [Count of Participants; unit: Participants]
  1 | 6 | 5 | 2 | 13
  ≤ 5 | 9 | 8 | 7 | 24
  ≥5 | 4 | 1 | 1 | 6
  No | 13 | 18 | 22 | 53
ACLS/BLS certification [Count of Participants; unit: Participants]
  Yes | 24 | 30 | 28 | 82
  No | 8 | 2 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Team Performance Observation Tool
Description: The assessment of the medical team's teamwork performance was conducted using the Team Performance Observation Tool, which includes a 23-item rating checklist. This checklist is divided into five categories: team structure (four items), leadership (six items), communication (four items), situation monitoring (five items), and mutual support (four items). Scores for each item range from 1 (Very Poor) to 5 (Excellent), resulting in a cumulative score between 23 and 115. A higher score indicates better teamwork performance.
Time Frame: Pretest at the 0 week, posttest right after intervention at the 4 weeks, and follow-up test at the 16 weeks.
Population: The total number of participants was 124, with 28 did not complete the pretest, resulting in 96 people completed pretest, intervention and posttest. Subsequently, 48 participants did not complete three-months follow up test , the total number of participants who completed the whole course reduced to 48. For participants who did not complete the study, the reasons included scheduling conflicts, staffing shortages in clinical settings, and surge in COVID-19 outbreak.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Board Game-based Learning | Simulation-based Learning | Lecture-based Learning
Number analyzed (Participants) | 32 | 32 | 32
score on a scale
  Pretest | 53.00 [47.00 to 59.00] | 39.00 [37.63 to 48.50] | 39.25 [35.75 to 53.50]
  Posttest | 57.75 [53.38 to 62.13] | 56.50 [49.63 to 59.88] | 51.50 [46.88 to 65.00]
  Three months follow-up: number analyzed (Participants) | 16 | 16 | 16
  Three months follow-up | 62.50 [46.63 to 67.50] | 56.75 [44.38 to 62.75] | 57.25 [49.13 to 68.00]
Statistical Analysis 1: Comparison: Board Game-based Learning vs Simulation-based Learning; For the pretest at week 0; Test type: Superiority; p < 0.05, Kruskal-Wallis; Median Difference (Final Values) = 12.75
Statistical Analysis 2: Comparison: Board Game-based Learning vs Simulation-based Learning; For posttest right after intervention at the 4 weeks; Test type: Superiority; p = 0.05, Kruskal-Wallis; Median Difference (Final Values) = 2.00
Statistical Analysis 3: Comparison: Board Game-based Learning vs Simulation-based Learning; For follow-up test at the 16 weeks; Test type: Superiority; p = 0.05, Kruskal-Wallis; Median Difference (Final Values) = 6.00

2. Primary Outcome: Knowledge of Teamwork Assessment
Description: The "Knowledge of Teamwork" assessment, aimed at evaluating healthcare professionals' understanding of teamwork knowledge, consists of 23 multiple-choice items based on the Team Strategies and Tools to Enhance Performance and Patient Safety (TeamSTEPPS) Learning Benchmarks provided by the Agency for Healthcare Research and Quality. Each item is formulated as a statement that participants must evaluate as true or false, choosing from five available answer options, of which only one is correct. Participants earn one point for each correct response, with no points awarded for incorrect answers, resulting in a total possible score of 0 to 23. A higher score signifies a more comprehensive understanding of the principles of teamwork knowledge.
Time Frame: Pretest at the 0 week, posttest right after intervention at the 4 weeks, and follow-up test at the 16 weeks.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Board-game Based Learning | Simulation-based Learning | Lecture-based Learning
Number analyzed (Participants) | 32 | 32 | 32
score on a scale
  Pretest | 18.00 [16.00 to 19.00] | 17.00 [16.00 to 19.00] | 17.00 [15.25 to 19.75]
  Posttest: number analyzed (Participants) | 32 | 32 | 30
  Posttest | 19.00 [17.00 to 20.00] | 18.00 [16.00 to 19.00] | 20.00 [17.00 to 21.00]
  Three months follow-up: number analyzed (Participants) | 16 | 16 | 16
  Three months follow-up | 19.00 [17.25 to 19.75] | 19.00 [18.00 to 19.95] | 19.50 [16.00 to 20.00]
Statistical Analysis 1: Comparison: Board-game Based Learning vs Simulation-based Learning; For pretest at the 0 week; Test type: Superiority; p < 0.05, Kruskal-Wallis; Median Difference (Final Values) = 1.00
Statistical Analysis 2: Comparison: Board-game Based Learning vs Simulation-based Learning; For posttest right after intervention at the 4 weeks; Test type: Superiority; p = 0.05, Kruskal-Wallis; Median Difference (Final Values) = 0.00
Statistical Analysis 3: Comparison: Board-game Based Learning vs Simulation-based Learning; For follow-up test at the 16 weeks; Test type: Superiority; p = 0.05, Kruskal-Wallis; Median Difference (Final Values) = 0.00

3. Secondary Outcome: Interprofessional Collaboration Scale
Description: The attitudes of healthcare professionals toward interprofessional collaboration were assessed using the 'Interprofessional Collaboration Scale' (IPC), which consists of 26 items. The Interprofessional Collaboration Scale covers three main aspects: communication, accommodation, and isolation. We adopted the first 13 items because they are relevant to medical and nursing professional backgrounds. The scale ranges from 1 (strongly disagree) to 4 (strongly agree), with total scores ranging from 13 to 52. A higher score indicates a more positive attitude toward interprofessional collaboration.
Time Frame: Pretest at the 0 week, posttest right after intervention at the 4 weeks, and follow-up test at the 16 weeks.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Board-game Based Learning | Simulation-based Learning | Lecture-based Learning
Number analyzed (Participants) | 32 | 32 | 32
score on a scale
  Pretest: number analyzed (Participants) | 32 | 31 | 32
  Pretest | 36.00 [35.00 to 41.00] | 40.00 [36.00 to 46.00] | 38.00 [36.00 to 41.00]
  Posttest: number analyzed (Participants) | 32 | 32 | 30
  Posttest | 41.00 [37.50 to 45.00] | 45.00 [38.00 to 50.00] | 39.00 [37.00 to 45.50]
  Three months follow-up: number analyzed (Participants) | 16 | 15 | 16
  Three months follow-up | 40.00 [39.00 to 47.75] | 43.00 [37.00 to 50.00] | 38.50 [37.00 to 48.25]
Statistical Analysis 1: Comparison: Board-game Based Learning vs Simulation-based Learning; For the pretest at week 0; Test type: Superiority; p < 0.05, Kruskal-Wallis; Median Difference (Final Values) = 40.00
Statistical Analysis 2: Comparison: Board-game Based Learning vs Simulation-based Learning; For posttest right after intervention at the 4 weeks; Test type: Superiority; p = 0.05, Kruskal-Wallis; Median Difference (Final Values) = 45.00
Statistical Analysis 3: Comparison: Board-game Based Learning vs Simulation-based Learning; For follow-up test at the 16 weeks; Test type: Superiority; p = 0.05, Kruskal-Wallis; Median Difference (Final Values) = 43.00

4. Secondary Outcome: Resuscitation Knowledge Scale
Description: The healthcare professionals' resuscitation medical knowledge was assessed using the 'Adavance Cardiac Life Support Precourse Self-Assessment,' which consisted of 60 items. The assessment covered three main aspects: rhythm identification, pharmacology, and practical application. We selected 20 items related to resuscitation medical management (ventricular tachycardia, ventricular fibrilation, asystole, pulseless electrical activity). The total score ranged from 0 (minimum) to 20 (maximum), with higher scores indicating a better understanding of resuscitation medical knowledge.
Time Frame: Pretest at the 0 week, posttest right after intervention at the 4 weeks, and follow-up test at the 16 weeks.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Board-game Based Learning | Simulation-based Learning | Lecture-based Learning
Number analyzed (Participants) | 32 | 32 | 32
score on a scale
  Pretest | 7.00 [5.25 to 10.00] | 8.00 [6.00 to 9.00] | 7.00 [5.25 to 10.50]
  Posttest: number analyzed (Participants) | 32 | 32 | 31
  Posttest | 11.00 [8.00 to 13.00] | 11.00 [8.25 to 13.00] | 11.00 [8.00 to 13.00]
  Three months follow-up: number analyzed (Participants) | 16 | 16 | 16
  Three months follow-up | 8.50 [6.25 to 10.00] | 7.00 [5.25 to 10.00] | 7.50 [6.25 to 10.75]
Statistical Analysis 1: Comparison: Board-game Based Learning vs Simulation-based Learning; For the pretest at week 0; Test type: Superiority; p < 0.05, Kruskal-Wallis; Median Difference (Final Values) = 0.00
Statistical Analysis 2: Comparison: Board-game Based Learning vs Simulation-based Learning; For posttest right after intervention at the 4 weeks; Test type: Superiority; p = 0.05, Kruskal-Wallis; Median Difference (Final Values) = 0.00
Statistical Analysis 3: Comparison: Board-game Based Learning vs Simulation-based Learning; For follow-up test at the 16 weeks; Test type: Superiority; p = 0.05, Kruskal-Wallis; Median Difference (Final Values) = 2.50

5. Secondary Outcome: Medical Task Performance
Description: The medical team's resuscitation management performance was assessed using the "Medical Task Performance" checklist. The checklist items were referenced from the 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Twenty items were identified by an expert panel based on the resuscitation guidelines, including applying adequate oxygen according to the patient's dynamic condition, timely identification of cardiac arrest and provision of high-quality cardiopulmonary resuscitation, identification of shockable rhythms and delivery of timely and correct shocks, and correct administration of resuscitation medication. The checklist was rated on a dichotomous scale with scores of 2 (complete), 1 (partial), and 0 (incomplete). The total score ranged from 0 (minimum) to 40 (maximum), with higher scores indicating better resuscitation management performance by the medical team.
Time Frame: Pretest at the 0 week, posttest right after intervention at the 4 weeks, and follow-up test at the 16 weeks.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Board-game Based Learning: The team of PGY doctors and nurses received training in resuscitation teamwork skills through a board-game based learning approach.
Arm/Group | Board-game Based Learning | Simulation-based Learning | Lecture-based Learning
Number analyzed (Participants) | 32 | 32 | 32
score on a scale
  Pretest | 23.00 [16.38 to 25.38] | 13.25 [10.75 to 17.75] | 22.00 [15.38 to 28.25]
  Posttest | 29.00 [25.13 to 31.38] | 27.25 [24.88 to 30.75] | 27.00 [23.38 to 32.25]
  Three months follow-up: number analyzed (Participants) | 16 | 16 | 16
  Three months follow-up | 29.25 [21.13 to 30.63] | 28.50 [23.25 to 30.75] | 22.00 [13.25 to 34.88]
Statistical Analysis 1: Comparison: Board-game Based Learning vs Simulation-based Learning; For the pretest at week 0; Test type: Superiority; p < 0.05, Kruskal-Wallis; Median Difference (Final Values) = 6.75
Statistical Analysis 2: Comparison: Board-game Based Learning vs Simulation-based Learning; For posttest right after intervention at the 4 weeks; Test type: Superiority; p = 0.05, Kruskal-Wallis; Median Difference (Final Values) = 0.25
Statistical Analysis 3: Comparison: Board-game Based Learning vs Simulation-based Learning; For follow-up test at the 16 weeks; Test type: Superiority; p = 0.05, Kruskal-Wallis; Median Difference (Final Values) = 0.00

6. Secondary Outcome: Learning Cognitive Load
Description: The learning cognitive load of healthcare professionals was assessed using the 'Chinese Version of the Learning Cognitive Load Questionnaire,' which consists of 8 items. The questionnaire encompasses two main aspects: mental load and mental effort. The scale ranges from 1 (Strongly Disagree) to 6 (Strongly Agree), with a total score from 6 (minimun) to 48 (maximun). A higher score indicates a higher learning cognitive load.
Time Frame: The posttest right after intervention at the 4 weeks.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Board-game Based Learning | Simulation-based Learning | Lecture-based Learning
Number analyzed (Participants) | 32 | 32 | 31
score on a scale | 22.00 [16.50 to 28.50] | 22.00 [15.25 to 27.00] | 21.00 [16.00 to 28.00]
Statistical Analysis 1: Comparison: Board-game Based Learning vs Simulation-based Learning; For posttest right after intervention at the 4 weeks; Test type: Superiority; p < 0.05, Kruskal-Wallis; Median Difference (Final Values) = 22.00

ADVERSE EVENTS:
Time Frame: Pretest at the 0 week, posttest right after intervention at the 4 weeks, and follow-up test at the 16 weeks.
Description: The study focused on assessing learning effectiveness, using educational procedures as both the assessment and intervention, without involving any invasive medical procedures or medical treatment. In the Adverse Event Reporting, regarding the monitoring/assessment of all-cause mortality, serious, or other (non-serious) adverse events, none of the participants experienced any adverse events throughout the study.
Groups:
- Board-game Based Learning: The team of PGY doctors and nurses, including total 32 participants, received 3 hours training intervention in resuscitation teamwork skills through a board game-based teaching approach. The intervention itself is an educational procedure, which is not including a medical treatment.
- Simulation-based Learning: The team of PGY doctors and nurses, including total 32 participants, received 3 hours training intervention in resuscitation teamwork skills through a simulation-based teaching approach. The intervention itself is an educational procedure, which is not including a medical treatment.
- Lecture-based Learning: The team of PGY doctors and nurses, including total 32 participants, received 3 hours training intervention in resuscitation teamwork skills through a interactive lecture-based learning approach. The intervention itself is an educational procedure, which is not including a medical treatment.
Arm/Group | Board-game Based Learning | Simulation-based Learning | Lecture-based Learning
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT05302414/Prot_SAP_000.pdf